CLINICAL TRIAL: NCT04234373
Title: Understanding Gut-brain Interactions and the Effect of a Low-carb Dietary Intervention in Obese Patients With and Without Glucose Intolerance or Diabetes: a Pilot Trial
Brief Title: Effect of a Low-carb Dietary Intervention in Obese Patients: a Pilot Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCP Obese
Record Dates: First submitted 2020-01-09; First posted 2020-01-21 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Glucose Intolerance; Obesity
MeSH Terms: conditions — Glucose Intolerance; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Carb dietary Intervention (Experimental)
  Interventions: Other: Low Carb diet

INTERVENTIONS:
Other: Low Carb diet — Low Carb diet (max. 130g carbohydrates/d) for 6 months

SUMMARY:
Effects of a 6 months low-carb dietary intervention on glycemic control, body composition and gut-brain interaction in obese and lean patients with and without glucose intolerance or diabetes

ELIGIBILITY:
Inclusion Criteria:

Group A: HEALTHY LEAN CONTROLS

* Healthy normal weight subjects with a body-mass index of 19.0-24.9kg/m2, HbA1C <5.7% and fasting glucose <5.6 mmol/l
* Normal eating habits
* Stable body weight for at least three months
* Informed Consent as documented by signature

Group B: PRE-DIABETIC or DIABETIC OBESE

* Pre-diabetic/Diabetic obese with a HbA1C >5.7% and/or fasting glucose >5.6 mmol/l) and body-mass index > 30kg/m2, otherwise healthy
* Normal eating habits
* Stable body weight for at least three months
* Informed Consent as documented by signature

Exclusion Criteria:

Group A: HEALTHY LEAN CONTROLS

* Pre-existing low carb diet (less than 45% of daily energy intake by carbohydrates)
* Pre-existing diet (vegetarian, vegan, gluten-free etc.)
* Psychiatric illness
* Alcohol abuse, (smoking allowed)
* Regular intake of medications, (oral contraceptives allowed)
* Intake of antibiotics within the last 3 months before inclusion
* Regular intake of pro- or prebiotics
* Chronic diseases of the gastrointestinal tract, history of gastrointestinal surgery with major changes to the gastrointestinal tract (e.g. bariatric surgery)
* Clinically relevant acute or chronic inflammatory disease
* Pregnancy
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Group B: PRE-DIABETIC or DIABETIC OBESE

* Pre-existing low carb diet (less than 45% of daily energy intake by carbohydrates)
* Pre-existing diet (vegetarian, vegan, gluten-free etc.)
* Psychiatric illness
* Alcohol abuse, (smoking allowed)
* Regular intake of medications (except: oral contraceptives, metformin, SGLT-2, statins, and antihypertensive, which are allowed)
* Intake of antibiotics within the last 3 months before inclusion
* Regular intake of pro- or prebiotics
* Chronic diseases of the gastrointestinal tract, history of gastrointestinal surgery with major changes to the gastrointestinal tract (e.g. bariatric surgery)
* Clinically relevant acute or chronic inflammatory disease
* Pregnancy
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Effect of a low-carb dietary intervention on glycemic control as defined by blood glucose level at 2h after an oral glucose tolerance test. | Change from baseline to 6 months

SECONDARY OUTCOMES:
Effect of a low-carb dietary intervention on body composition as measured with dual-energy x-ray absorptiometry | Change from baseline to 6 months
Effect of a low-carb dietary intervention on metabolomics as measured in plasma, urine and stool samples | Change from baseline to 6 months
  Metabolomic analysis of the bacterial metabolites present in the urine by combining nuclear magnetic resonance (1H-NMR) and mass spectrometry
Effect of a low-carb dietary intervention on gut microbiota composition as measured in stool samples | Change from baseline to 6 months
  Human gut microbiota composition measured with metagenomic shotgun sequencing
Effect of a low-carb dietary Intervention on brain network activity as measured with functional MRI | Change from baseline to 6 months
Effect of a low-carb dietary intervention on liver fat fraction as measured with MRI | Change from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Wölnerhanssen, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- St Clara Research Ltd, St Claraspital Basel, Basel, Switzerland